CLINICAL TRIAL: NCT06297304
Title: Determining the Influence of an Intervention Based on Sedentary Behavior Reduction and Physical Activity Promotion Among Medical Students.
Brief Title: Sedentary Behaviors Reduction and Physical Activity Promotion for Optimal Medical StudentS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Research on Healthcare Performance Lab U1290 (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: PROMESS - PHYSICAL ACTIVITY
Record Dates: First submitted 2024-02-29; First posted 2024-03-07 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Health Behavior; Health-Related Behavior; Physical Inactivity; Sedentary Behavior; Sedentary Time
Keywords: Health; Student; Curriculum; Behaviour; Medical; Physical activity; Sedentary
MeSH Terms: conditions — Health Behavior; Sedentary Behavior; Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: All volunteers will receive a physical activity and sedentary management intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical Activity Intervention (Experimental): One arm : all volunteers will receive an intervention program based on sedentary behavior reduction and physical activity promotion.
  Interventions: Behavioral: Sedentary and physical activity behaviors

INTERVENTIONS:
Behavioral: Sedentary and physical activity behaviors — The intervention will consist of three individual sessions, each lasting one hour, with approximately 15 days between each session. The sessions will be scheduled as follow: Week 5 and 6 (session 1), week 7 and 8 (session 2), week 9, 10, and 11 (session 3). During these sessions, subjective and objective indicators related to sedentary behaviors and the physical activity levels will be recorded to assess the progress of each student.

SUMMARY:
Medical students are under great competitive pressure throughout their studies. Our field surveys conducted in 2022 and 2023 at the Lyon Est Faculty of Medicine revealed that 78% of 482 students showed an excessive sedentary lifestyle compared to the threshold set by WHO. It is expected that a low level of physical activity and/or too high a sedentary lifestyle deteriorates significantly their quality of life and their health. In 2014, a British survey of 356 students in Medicine showed that lack of physical activity was an major predictor of burnout symptoms. Numerous studies show that regular physical activity improves the mental health of students and their cognitive performance.

The PROMESS - PHYSICAL ACTIVITY project aims to offer solutions to students to decrease their sedentary behavior and to improve their physical activity level during their medical studies through an intervention program. From a long term perspective, this intervention may also prevent disorders related to inadequate levels of physical activity and/or sedentary behavior. It responds to a demand expressed by students : our previous field study showed that 45% of fourth-year students declared being "very interested and/or interested" in following an intervention that aimed at improving physical activity. The objective of this study is to determine the influence of an intervention based on sedentary behavior reduction and physical activity promotion among medical students.

DETAILED DESCRIPTION:
Our project aims to help future healthcare professionals to adopt health-promoting behaviors during their studies in a preventive approach. This support will be provided through an intervention of physical activity management during their curriculum. Specifically, 4th and 5th-year students at the Faculty of Medicine of Lyon Est will have the opportunity to participate in the PROMESS PHYSICAL ACTIVITY project. This intervention will span 11 weeks. At the end of this period, we expect improvements in both subjective and objective indicators of physical activity and sedentary.

METHODS.

PRE-INTERVENTION. Week 1-3. Students will undergo a two-hour session, during which, they will complete questionnaires on physical activity and sedentary behavior. Bioimpedance measurements will be recorded. Students will also perform three physical fitness tests (vertical jump, maximal isometric strength and endurance). Then, they will wore actimeters to record sedentary behaviors and physical activity levels during three weeks (from week 1 to week 3).

INTERVENTION. From week 5 to week 11. The intervention will consist of three individual sessions, each lasting one hour, with approximately 15 days between each session. Each session includes individual interview between a physical activity expert and the participant (i.e. student).The sessions will be scheduled as follow: week 5 and 6 (session 1), week 7 and 8 (session 2), week 9, 10, and 11 (session 3). During the interview, the expert will realize an initial assessment of student physical activity and sedentary behavior levels and will give personalized goals to student. Subsequent sessions will follow the same structure.

ELIGIBILITY:
Inclusion Criteria:

* Being a 4th-year or a 5th-year medical student at the Faculty of Medicine Lyon East during the academic year 2023-2024.
* Having read the information note.
* Having signed the written consent.

Exclusion Criteria:

-No exclusion criteria will be applied.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-11-11 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Perceived level of sedentary : Evolution of the score obtained at the Rapid Physical Activity Questionnaire (RPAQ) on sedentary behaviors. | From week 5 to week 11.
  The students level of sedentary behaviors will be assessed through the RPAQ questionnaire.This questionnaire includes questions about sedentary behaviors, such as time spent sitting down.Scores are expressed in hours per day for week and weekend days. The measure will be done every session, i.e. session 1 (week 5-6), session 2 (week 7-8) and session 3 (week 9,10,11).

SECONDARY OUTCOMES:
Perceived level of physical activity : Score obtained at the Global Physical Activity Questionnaire (GPAQ) on physical activity levels. | Week 1 (Pre-intervention)
  The students basal level of physical activity will be assessed through the GPAQ questionnaire. Scores are expressed in MET.min week. It can be divided into six sub-scores (i.e level of moderate and intense physical activity, physical activity during leisure activity, physical activity during locomotion, physical activity at work and sedentarity levels). This measure will be done during the pre-interventional period at week 1.
Perceived level of sedentary : Score obtained at the Rapid Physical Activity Questionnaire (RPAQ) on sedentary behaviors. | Week 1 (Pre-intervention)
  The students basal level of sedentary behavior will be assessed through the RPAQ questionnaire.This questionnaire typically includes questions about sedentary behaviors, such as time spent sitting down. Scores are expressed in hours per day. This measure will be done during the pre-interventional period at week 1.
Actimetry records.Total activity during the pre-intervention. | From week 1 to week 3 (pre-intervention).
  The objective students levels of physical activity and sedentary behavior will be accessed through the actimetry recordings.The total activity time represents the total duration of physical activity within the monitoring period, measured in hours.The measure will be done in continuous from week 1 to week 3 (pre-intervention).
Actimetry records. Moderate-to-vigorous Physical Activity (MVPA) during the pre-intervention. | From week 1 to week 3 (pre-intervention).
  The objective students levels of physical activity and sedentary behavior will be accessed through the actimetry recordings. Moderate-to-vigorous physical activity (MVPA) refers to physical activities that require moderate to high levels of effort and significantly increase heart rate and breathing. These activities contribute to improved cardiovascular health, fitness, and overall well-being. MVPA encompasses a range of activities that are more intense than sedentary behaviors but less intense than vigorous activities. MVPA is measured in minutes/day. The measure will be done in continuous from week 1 to week 3 (pre-intervention).
Actimetry records. Light Physical Activity during the pre-intervention. | From week 1 to week 3 (pre-intervention).
  The objective students levels of physical activity and sedentary behavior will be accessed through the actimetry recordings. Light physical activity refers to any activity that requires minimal effort and only slightly elevated heart rate and breathing, measured in minutes/day. It involves movement that is more than sedentary behavior but does not reach the intensity level of moderate-to-vigorous physical activity (MVPA). Light physical activities are typically those that can be performed during daily tasks or leisurely pursuits and do not typically lead to significant sweating or increased breathing rate.The measure will be done in continuous from week 1 to week 3 (pre-intervention).
Actimetry records. Steps count during the pre-intervention. | From week 1 to week 3 (pre-intervention).
  The objective students levels of physical activity and sedentary behavior will be accessed through the actimetry recordings.The total number of steps count per day during the monitoring period, which provides a measure of ambulatory activity. The measure will be done in continuous from week 1 to week 3 (pre-intervention).
Actimetry records. Energy expenditure during the pre-intervention. | From week 1 to week 3 (pre-intervention).
  The objective students levels of physical activity and sedentary behavior will be accessed through the actimetry recordings. Energy expenditure refers to the amount of energy, measured in calories or joules, that an individual uses or expands during a specific period of time. The measure will be done in continuous from week 1 to week 3 (pre-intervention).
Actimetry records. Number of sedentary breaks during the pre-intervention. | From week 1 to week 3 (pre-intervention).
  The objective students levels of physical activity and sedentary behavior will be accessed through the actimetry recordings. Sedentary breaks refer to short periods of time during which individuals interrupt prolonged sitting or sedentary behavior by engaging in light physical activity or standing. The measure will be done in continuous from week 1 to week 3 (pre-intervention).
Actimetry records. Sedentary time during the pre-intervention. | From week 1 to week 3 (pre-intervention).
  The objective students levels of physical activity and sedentary behavior will be accessed through the actimetry recordings. The sedentary time is the total duration of sedentary behavior, defined as periods of minimal movement or activity, measured in minutes/day. The measure will be done in continuous from week 1 to week 3 (pre-intervention).
Actimetry records. Number of prolonged sedentary bouts during the pre-intervention. | From week 1 to week 3 (pre-intervention).
  The objective students levels of physical activity and sedentary behavior will be accessed through the actimetry recordings. Prolonged sedentary bouts refer to extended periods of time during which individuals engage in minimal physical activity or remain in a seated or reclined position without interruption. These bouts typically last for prolonged durations, measured in minutes/day, often exceeding 30 minutes or more at a time.The measure will be done in continuous from week 1 to week 3 (pre-intervention).
Actimetry records.Vector of the dynamic body acceleration (VeDBA) during the pre-intervention. | From week 1 to week 3 (pre-intervention).
  The objective students levels of physical activity and sedentary behavior will be accessed through the actimetry recordings. The vector of the dynamic body acceleration (VeDBA) quantifies the dynamic acceleration of an body movements in three-dimensional space. The dynamic acceleration captured by the accelerometer reflects the intensity, accounting for both changes in speed and changes in direction. Researchers use VeDBA as a proxy for overall energy expenditure or activity levels in natural environments. Higher VeDBA values typically indicate more vigorous or energetic movements, while lower values suggest periods of rest or low activity. The measure will be done in continuous from week 1 to week 3 (pre-intervention).
Body composition markers. Body Mass Index (BMI) during the pre-intervention. | Week 1 (Pre-intervention)
  The Body Mass Index (BMI) is a measure used to assess an individual's body weight in relation to their height. It's calculated by dividing a person's weight in kilograms by the square of their height in meters (BMI = weight in kilograms / (height in meters)²). BMI provides a general indication of whether a person's weight falls within a healthy range relative to their height. Here's how BMI categories are typically interpreted:
  Underweight: BMI less than 18.5 Normal weight: BMI between 18.5 and 24.9 Overweight: BMI between 25 and 29.9 Obesity: BMI 30 or greater. The measure will be done at week 1 (pre-intervention).
Body composition markers. Skeletal muscle mass measured by bioimpedancemetry during the pre-intervention. | Week 1 (Pre-intervention)
  The students body composition will be assessed using impedance metric variables. Skeletal muscle mass refers to the total mass or amount of skeletal muscle tissue in the body. It's often expressed in kilograms or as a percentage of total body weight.The measure will be done at week 1 (pre-intervention).
Body composition markers. Fat mass measured by bioimpedancemetry during the pre-intervention. | Week 1 (Pre-intervention)
  The students body composition will be assessed using impedance metric variables.The fat mass metric represents the total amount of body fat. It's often expressed in kilograms or as a percentage of total body weight. The measure will be done at week 1 (pre-intervention).
Body composition markers. Total body hydration measured by bioimpedancemetry during the pre-intervention. | Week 1 (Pre-intervention)
  The students body composition will be assessed using impedance metric variables.The total body hydration metric represents the total amount of water present in the body, including intracellular and extracellular water compartments. It's often expressed in liters or as a percentage of total body weight. The measure will be done at week 1 (pre-intervention).
Physical Fitness markers - Strength. The force developed during a maximal isometric contraction of the quadriceps during the pre-intervention. | Week 1 (Pre-intervention)
  The students basal level of physical fitness will be assessed through a muscular strength test. The measure will be done at week 1 (pre-intervention).
Physical Fitness markers markers - Power. Height of jump during the pre-intervention. | Week 1 (Pre-intervention)
  The students basal level of physical fitness will be assessed through a power test, a vertical jump.
  The squat jump is plyometric exercise in which a person bends their knees to lower their body into a squat position, then performs an explosive jump upwards by extending the hips, knees, and ankles simultaneously. During this exercise, the height of jump will be measured. The measure will be done at week 1 (pre-intervention).
Physical Fitness markers - Power. Time of flight during the pre-intervention. | Week 1 (Pre-intervention)
  The students basal level of physical fitness will be assessed through a power test, a vertical jump. During this exercise, the time of flight will be measured. The measure will be done at week 1 (pre-intervention).
Physical Fitness markers - Power. Relative Power during the pre-intervention. | Week 1 (Pre-intervention)
  The students basal level of physical fitness will be assessed through a power test, a vertical jump. During this exercise, the relative power can be estimated. The measure will be done at week 1 (pre-intervention).
Physical Fitness markers - Endurance. Speed through the endurance test during the pre-intervention. | Week 1 (Pre-intervention)
  The students basal level of physical fitness will be assessed through a cardiorespiratory endurance test (modified VAMEVAL). The measure will be done at week 1 (pre-intervention).
Physical Fitness markers - Endurance. VO2max through the endurance test during the pre-intervention. | Week 1 (Pre-intervention)
  The students basal level of physical fitness will be assessed through a cardiorespiratory endurance test (modified VAMEVAL).
  During this test, the velocity at maximal aerobic (VMA) is the maximum speed (velocity) reached where the individual can still maintain aerobic metabolism without transitioning into anaerobic metabolism. VO2max refers to the maximum rate of oxygen consumption during intense exercise, typically measured in milliliters of oxygen per kilogram of body weight per minute (ml/kg/min). It is a key indicator of an individual's cardiovascular fitness and aerobic endurance. The VO2max was estimated as 3.5 times VMA. The measure will be done at week 1 (pre-intervention).
Physical Fitness markers - Endurance. Heart rate during the endurance test during the pre-intervention. | Week 1 (Pre-intervention)
  The students basal level of physical fitness will be assessed through a cardiorespiratory endurance test (modified VAMEVAL). The heart rate will be measured at three moments: maximum, submaximal, at 1 minute, and 3 minutes of recovery. The measure will be done at week 1 (pre-intervention).
Perceived level of physical activity : Evolution of the score obtained at the Global Physical Activity Questionnaire (GPAQ) on physical activity level. | From week 5 to week 11.
  The students level of physical activity will be assessed through the GPAQ questionnaire. Scores are expressed in MET.min week. It can be divided into six sub-scores (i.e level of moderate and intense physical activity, physical activity during leisure activity, physical activity for locomotion, physical activity at work locomotion and sedentarity level). The measure will be done every session, i.e. session 1 (week 5-6), session 2 (week 7-8) and session 3 (week 9,10,11).
Actimetry records. Evolution in Total activity during the intervention. | From week 5 to week 11.
  The measure will be done between every session, i.e. between session 1 (week 5-6) and session 2 (week 7-8) and between session 2 and session 3 (week 9,10,11).
Actimetry records. Evolution in Moderate-to-vigorous physical activity (MVPA) during the intervention. | From week 5 to week 11.
  The measure will be done between every session, i.e. between session 1 (week 5-6) and session 2 (week 7-8) and between session 2 and session 3 (week 9,10,11).
Actimetry records. Evolution in Light physical activity measured in min/day during the intervention. | From week 5 to week 11.
  The measure will be done between every session, i.e. between session 1 (week 5-6) and session 2 (week 7-8) and between session 2 and session 3 (week 9,10,11).
Actimetry records. Evolution in Step Count during the intervention. | From week 5 to week 11.
  The measure will be done between every session, i.e. between session 1 (week 5-6) and session 2 (week 7-8) and between session 2 and session 3 (week 9,10,11).
Actimetry records. Evolution in Energy expenditure during the intervention. | From week 5 to week 11.
  The measure will be done between every session, i.e. between session 1 (week 5-6) and session 2 (week 7-8) and between session 2 and session 3 (week 9,10,11).
Actimetry records. Evolution in number of sedentary breaks during the intervention. | From week 5 to week 11.
  The measure will be done between every session, i.e. between session 1 (week 5-6) and session 2 (week 7-8) and between session 2 and session 3 (week 9,10,11).
Actimetry records. Evolution in Number of prolonged sedentary bouts during the intervention. | From week 5 to week 11.
  The measure will be done between every session, i.e. between session 1 (week 5-6) and session 2 (week 7-8) and between session 2 and session 3 (week 9,10,11).
Actimetry records. Evolution in the vector of the dynamic body acceleration (VeDBA) during the intervention. | From week 5 to week 11.
  The measure will be done between every session, i.e. between session 1 (week 5-6) and session 2 (week 7-8) and between session 2 and session 3 (week 9,10,11).
Body composition markers. Evolution in BMI during the intervention. | From week 5 to week 11.
  The measure will be done every session, i.e. session 1 (week 5-6), session 2 (week 7-8) and session 3 (week 9,10,11).
Body composition markers. Evolution in fat mass measured by bioimpedancemetry during the intervention. | From week 5 to week 11.
  The measure will be done every session, i.e. session 1 (week 5-6), session 2 (week 7-8) and session 3 (week 9,10,11).
Body composition markers: Impedance metric measures. Evolution in skeletal muscle mass measured by bioimpedancemetry during the intervention. | From week 5 to week 11.
  The measure will be done every session, i.e. session 1 (week 5-6), session 2 (week 7-8) and session 3 (week 9,10,11).
Body composition markers: Impedance metric measures. Evolution in total body hydration measured by bioimpedancemetry during the intervention. | From week 5 to week 11.
  The measure will be done every session, i.e. session 1 (week 5-6), session 2 (week 7-8) and session 3 (week 9,10,11).
VAS - physical fitness: Evolution of the score obtained at the 100-mm Visual Analogue Scale (VAS) assessing the perceived level of physical fitness. | From week 5 to week 11.
  The students level of physical fitness will be assessed on a 100-mm Visual Analogue Scale (VAS: "Over the past two weeks, how would you characterize your level of physical fitness?") ranging from 0 (bad shape) to 100 (best shape ever). The measure will be done every session, i.e. session 1 (week 5-6), session 2 (week 7-8) and session 3 (week 9,10,11).
VAS - physical activity. Evolution of the score obtained at the 100-mm Visual Analogue Scale (VAS) assessing the perceived level of physical activity. | From week 5 to week 11.
  The students level of physical activity will be assessed on a 100-mm Visual Analogue Scale (VAS: "Over the past two weeks, how would you characterize your level of physical activity?") ranging from 0 (completely inactive) to 100 (extremely active).The measure will be done every session, i.e. session 1 (week 5-6), session 2 (week 7-8) and session 3 (week 9,10,11).
VAS - sedentary behaviours. Evolution of the scores obtained at the 100-mm Visual Analogue Scale (VAS) assessing the perceived level of sedentary behaviours. | From week 5 to week 11.
  The students level of sedentary behaviours will be assessed on a 100-mm Visual Analogue Scale (VAS: "Over the past two weeks, how would you characterize your level of sedentary behaviours?") ranging from 0 (extremely sedentary) to 100 (absolutely not sedentary). The measure will be done every session, i.e. session 1 (week 5-6), session 2 (week 7-8) and session 3 (week 9,10,11).
Advices given by the expert. Score obtained on a Likert scale ranging from 1 to 5 characterizing the nature of the advices given by the expert. | From week 5 to week 11.
  Following each session, the expert reported if he/she has given during the interview a specific advice according to a pre-established list. For each pre-established advice, he/she has to report if :
  1. He/she didn't mention this
  2. He/she mentioned this but didn't directly advise it
  3. He/she mentioned this and recommended it
  4. He/she had set this in the goals
  5. The student was already doing it (positive reinforcement). The measure will be done every session, i.e. session 1 (week 5-6), session 2 (week 7-8) and session 3 (week 9,10,11).
Likert - expert estimation of student's achievements. Score obtained on a Likert scale ranging from 1 to 3 accessing if the expert estimates that the student has achieve the goals previously set. | From week 7 to week 11.
  The expert evaluates, from 0 to 3 (i.e. 0 : not achieved at all, 1: slightly achieved, 2: fairly well achieved, 3: well achieved) if he/she estimates that the student has achieve the goals previously set.The measure will be done at session 2 (week 7-8) and session 3 (week 9,10,11).
Likert - expert satisfaction. Scores obtained on a Likert scale ranging from 1 to 5 accessing the expert's satisfaction of his/her intervention. | From week 5 to week 11.
  The perceived level of the expert satisfaction ("Are you satisfied with the session you just realized?") will be accessed on a likert scale ranging from 1 (not at all satisfied) to 5 (very satisfied). The measure will be done every session, i.e. session 1 (week 5-6), session 2 (week 7-8) and session 3 (week 9,10,11).
Likert - expert level of comfort. Score assessing the expert comfort levels in participant relationships on a likert scale ranging from 1 to 5. | From week 5 to week 11.
  The perceived level of expert comfort of the relationship with the student ("How comfortable did you feel with the student?") will be accessed on a likert scale ranging from 1 (not at all comfortable) to 5 (very comfortable). The measure will be done every session, i.e. session 1 (week 5-6), session 2 (week 7-8) and session 3 (week 9,10,11).
Likert - expert estimation of the overall student's achievements. Score obtained on a Likert scale ranging from 1 to 5 accessing the expert's level of satisfaction on the student's progress. | Week 9-10-11
  The level of expert satisfaction of the student's progress ("Are you satisfied with the student's progress during the all intervention?") will be accessed on a likert scale ranging from 1 (not at all satisfied) to 5 (very satisfied). This measure will be done at the session 3, i.e. approximately at week 9,11,10.
Composite score - Student's satisfaction. Score ranging from 0 to 100 accessing the student's level of satisfaction of the all intervention. | Week 9-10-11
  The composite score will be the mean of two sub-scores :
  1. An intervention specific score. Mean of the scores obtained at the three 100-mm Visual Analogue Scales ranging from 0 (absolutely not) to 100 (completely) :
     * VAS: "Do you think the module has helped you increase your level of physical fitness?")
     * VAS: "Do you think the module has helped you increase your level of physical activity?")
     * VAS: "Do you think the module has helped you decrease your level of sedentary behaviours?")
  2. An intervention general score. Mean of the scores obtained at the two 100-mm Visual Analogue Scales ranging from 0 (absolutely not) to 100 (completely) :
     * VAS :"Do you think the proposed goals were suitable for your daily life?"
     * VAS: "Do you think you can sustain the habit changes?"
  Theses measures will be done at the session 3, i.e. approximately at week 9,11,10.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Schlatter, Dr., Principal Investigator — RESHAPE U1290 INSERM UCBL-LYON 1 Rockfeller, Lyon France.
Locations (1):
- RESHAPE, Lyon, France